CLINICAL TRIAL: NCT06798792
Title: Evaluation of the Effect of Discharge Education Given With Two Different Teaching Techniques on Students' Self-Efficacy and Satisfaction Levels: A Randomized Trial
Brief Title: The Effect of Discharge Education Given With Two Different Teaching Techniques on Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Yağmur Kayın, Registered Nurse, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ykayin
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Nursing Students
Keywords: Nursing Education; Patient Education; Discharge Planning; Active Learning

STUDY DESIGN:
Intervention Model Description: A total of 180 students enrolled in the Surgical Diseases Nursing course at the Gülhane Faculty of Nursing, Health Sciences University were randomized into two groups based on their first-year cumulative academic grade point averages. The first group received Discharge Education using the PechaKucha technique, while the second group received it using the TeachBack technique.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A total of 180 nursing students enrolled in the 2nd-year Surgical Diseases Nursing course were randomized into two groups based on their 1st-year cumulative academic grade point average by an independent statistician, separate from the study and the data obtained was analyzed by a statistician who was independent of the study and not involved in its implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1. PechaKucha (Experimental): The students in Group 1 were taught the Discharge Education course using the PechaKucha teaching technique.
  PechaKucha, which translates to "chatter" or "chit-chat" in Japanese, was first introduced in 2003 in Tokyo within the field of architecture. It was initially used by architects to present new projects and structures and to exchange ideas. This method is a fast-paced, innovative teaching and presentation technique that consists of 20 slides, each containing minimal text and authentic visual metaphors. Each slide is displayed for 20 seconds using an automatic timer, making the total presentation 6 minutes and 40 seconds long.
  In Power Point presentations, this timing can be set by selecting the Transitions tab and adjusting the duration to 20 seconds for all slides. The goal of this method is to make presentations more dynamic, engaging, and enjoyable.
  Interventions: Other: PechaKucha technique
- Group 2. TeachBack (Experimental): The students in Group 2 were taught the Discharge Education course using the TeachBack teaching technique.
  The TeachBack method, also known as the "Tell Me What You Learned" technique, is a dynamic and interactive learning and teaching process. The primary goal of the TeachBack method is to ensure that the given education is correctly understood by having participants explain it back to the educator in their own words. If the purpose of the education is to teach a specific skill, the goal is to observe whether the learner can correctly perform the intended skill.
  This method helps eliminate communication barriers by allowing for immediate feedback on misunderstood or incomplete information while reinforcing correct knowledge. It serves as an effective teaching strategy to evaluate the extent of understanding, ensuring that learners fully grasp the subject matter.
  Interventions: Other: TeachBack technique

INTERVENTIONS:
Other: PechaKucha technique — The Discharge Education course was taught using the PechaKucha technique.
  Arms: Group 1. PechaKucha
Other: TeachBack technique — The Discharge Education course was taught using the TeachBack technique.
  Arms: Group 2. TeachBack

SUMMARY:
This study aims to examine the effects of PechaKucha and TeachBack teaching techniques, used in the instruction of the "Discharge Education" course for nursing students, on students' knowledge levels and self-efficacy regarding discharge education, as well as their satisfaction with the teaching method.

DETAILED DESCRIPTION:
The study was conducted as a randomized trial. Permission was obtained from the Gülhane Faculty of Nursing, Health Sciences University, and the Gülhane Scientific Research Ethics Committee, Health Sciences University. The study sample consisted of 180 students enrolled in the Surgical Diseases Nursing course at the Gülhane Faculty of Nursing, Health Sciences University, during the 2024-2025 Fall Semester. The students were randomized into two groups based on their first-year cumulative grade point averages. The first group received the "Discharge Education" course using the PechaKucha teaching technique, while the second group received it using the TeachBack teaching technique.

Data were collected using the Descriptive Characteristics Form, Discharge Education Knowledge Test, General Self-Efficacy Scale, and Adult Education Satisfaction Scale. Statistical analyses were performed using Shapiro-Wilk, Kolmogorov-Smirnov, and Mann-Whitney U tests, as well as Friedman Test Dunn-Bonferroni, Pearson Chi-Square, Fisher's Exact, and Fisher-Freeman-Halton tests. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd-year student at the Gülhane Faculty of Nursing, Saglık Bilimleri University
* Willing to participate in the study
* Being over 18 years old
* Taking the Surgical Diseases Nursing course for the first time

Exclusion Criteria:

* Wishing to withdraw from the study at any stage
* Incomplete completion of the data collection form related to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Self-efficacy level | The scale was administered to students before and after the Discharge Education course. It takes approximately 10 minutes to complete.
  To determine students' self-efficacy, the General Self-Efficacy Scale was used. This scale was developed by Sherer et al. (1982), and its Turkish validity and reliability study was conducted by Yıldırım and İlhan (2010). The scale follows a 5-point Likert format (1: Not at all, 5: Very well) and consists of 17 items. As the score obtained from the scale increases, general self-efficacy also increases. The minimum possible score is 17, while the maximum is 85. The internal consistency coefficient (Cronbach's alpha) of the scale was calculated as 0.80. Necessary permissions were obtained for the use of the General Self-Efficacy Scale.
Satisfaction level | The scale was administered to students after the completion of the Discharge Education course. It took approximately 10 minutes to complete.
  To determine students' satisfaction levels, the Adult Education Satisfaction Scale was used. This scale was developed and its validity and reliability study conducted by Yüksekbilgili et al. (2016). It consists of 30 items and includes six sub-dimensions: "Instructor's Presentation Skills, Instructor's Communication Skills, Learning Environment, Training Organization, Training Objectives, Training Outcomes, and General Evaluation."
  The scale uses a 5-point Likert format (1 = Strongly Disagree, 5 = Strongly Agree). As the score obtained from the scale increases, satisfaction levels also increase. The minimum possible score is 30, while the maximum is 150. The internal consistency coefficient (Cronbach's alpha) of the scale was calculated as 0.94. Necessary permissions were obtained before using the Adult Education Satisfaction Scale
Knowledge level | The test was administered to students before and after the Discharge Education course. It takes approximately 15 minutes to complete.
  To assess students' knowledge level regarding "Discharge Education," a multiple-choice test (with five options) consisting of 10 questions was developed by the researcher. The test is evaluated on a 100-point scale, with each correct answer worth 10 points.
  Before administering the Discharge Education Knowledge Test, expert opinions were obtained from five faculty members using the DAVIS method.

CONTACTS AND LOCATIONS:
Overall Officials: Yağmur Kayın, RN, Principal Investigator — Saglık Bilimleri University; Bediye Öztaş, Ph. D, Study Director — Saglık Bilimleri University
Locations (1):
- Saglık Bilimleri University, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No